CLINICAL TRIAL: NCT01353417
Title: A Single-site, Prospective Non-interventional-study With Adport Sandoz© Capsules for Prophylaxis of Graft Rejection in Patients With Stable Kidney Function After Renal Allograft.
Brief Title: Non-interventional-study With Tacrolimus Sandoz© Capsules for Prophylaxis of Renal Graft Rejection
Status: Completed | Type: Observational
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Other Study IDs: TAC SAN NIS 2011
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Insufficiency
Keywords: Grafting, kidney; Transplantation, kidney
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Retained types of biospecimen: whole blood, serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Renal allograft
  Interventions: Other: In this observational study no study specific intervention is planned

INTERVENTIONS:
Other: In this observational study no study specific intervention is planned — Patients with stable kidney function who already receive Tacrolimus Sandoz© capsules before being included in this non-interventional study, are being observed for 6 months by their attending physicians. Routine medical treatment is provided.

SUMMARY:
This non-interventional study intends to collect epidemiological data in patients with stable kidney function after renal transplantation, who receive Tacrolimus Sandoz© according to the approved indication.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18
* Post renal transplantation time: ≥ 6 months
* Stable kidney function ( serum creatinine < 3.0mg/dl; variation < 0.5mg/dl at 2 appointments in minimum distance of 6 days)
* Stable Tacrolimus Sandoz© dose > 2 weeks before inclusion in this Non Interventional Study (NIS)
* Written and oral informed consent

Exclusion Criteria:

* Well-known poor compliance with immunosuppressives
* Acute rejection reaction within the past 3 months or antibody-therapy because of rejection within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after renal transplantation who are treated in the general hospital of Vienna on an outpatient basis
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in Adport Sandoz© trough level | Observation time: 26 weeks

SECONDARY OUTCOMES:
Efficacy of Adport Sandoz© in prevention of renal graft rejection by observing serum creatinine levels | Observation time: 26 weeks
Incidence of serious adverse drug reactions | Observation time: 26 weeks
Incidence of adverse drug reactions | Observation time: 26 weeks
Incidence of serious adverse events | Observation time: 26weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital, Vienna, Austria